CLINICAL TRIAL: NCT04319419
Title: Effectiveness of a Supplement Containning Milk Proteins, Vitamins and Minerals to Reduce Fat Deposition, Systemic Inflammation and Improve Nutritional Status in Obese School-age Children
Brief Title: Milk Proteins and Micronutrient Supplementation in Obese Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Queretaro (Other)
Collaborators: NUCITEC S.A. de C.V. (Unknown)
Responsible Party: Principal Investigator, Jorge Luis Rosado Loria, Principal Investigator, Universidad Autonoma de Queretaro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNN201104
Record Dates: First submitted 2020-02-28; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Obesity, Childhood
Keywords: micronutrients; obesity; school-age children; milk proteins
MeSH Terms: conditions — Pediatric Obesity; Obesity | interventions — Micronutrients; Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Control group received only nutrition education and treated group received nutrition education plus a supplement with milk protein and micronutrients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement with micronutrients (Experimental): Nutrition education with a supplement
  Interventions: Dietary Supplement: Supplement with micronutrients
- Nutrition education (Experimental): Group received only nutrition education
  Interventions: Other: Nutrition education

INTERVENTIONS:
Dietary Supplement: Supplement with micronutrients — Obese children were divided in 2 groups. A group received the supplement plus nutrition education and other group was a control, only received nutrition education.
  Arms: Supplement with micronutrients
Other: Nutrition education — Group received nutrition education program during 6 months
  Arms: Nutrition education

SUMMARY:
Milk proteins and micronutrients could be beneficial in the prevention and treatment of obesity.

The objective was to evaluate a supplement with milk proteins and multivitamins and minerals with nutrition education on anthropometry, body composition, micronutrient status, blood pressure, lipid profile, systemic inflammation, leptin and insulin resistance in obese children at baseline and after 6 months.

DETAILED DESCRIPTION:
Obese children were selected in elementary schools from 5 rural communities of the State of Querétaro. One hundred fifty two obese children (Z-score >2 standard deviations) aged 6-11y were randomly assigned to receive one of two treatments: 1) 237mL/day of milk proteins and multiple micronutrients supplement (MPMS) plus Nutrition Education (NE) program or 2) NE alone for 24 weeks.

Children in both groups were evaluated at baseline and 6 months after treatment initiated. At both times the following variables were evaluated:

Visit 1 (Screening): Mothers and parents received oral and written information regarding all aspects of the study. Informed consent, medical history, demographic information, weight and height were obtained.

Visit 2 (Clinical Laboratory testing): A blood preasure and sample was taken by an specialist. Blood test included Glucose, total cholesterol, triglycerides, HDL cholesterol and LDL cholesterol, Tumor necrosis factor alpha (TNF-α), interleukin-6 (IL-6) and interleukin-10 (IL-10), C reactive protein, insulin and leptin.

Visit 3 (Nutrition Clinic at UAQ): body composition was determined by DEXA. The NE were given at Nutrition Clinic and school to the children's parents each week.

ELIGIBILITY:
Inclusion Criteria:

* Children with obesity (BMI>30)
* Aged: 6 to 11 years
* Both sex
* Parents accepted to participate and signed informant consent

Exclusion Criteria:

* Children with dyslipidemia
* Metabolic disease
* Hypertension
* Physical disability
* Using vitamins and minerals supplements and/or receiving treatment for obesity during the last 3 months.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 152 (Actual)
Dates: Start 2011-12-05 (Actual); Primary Completion 2012-12-05 (Actual); Study Completion 2012-12-05 (Actual)

PRIMARY OUTCOMES:
Total body fat | baseline to 6 months
  change in fat

SECONDARY OUTCOMES:
Total cholesterol | Beaseline to 6 months
  Change in total cholesterol
HDL | Baseline to 6 months
  change in HDL
LDL | baseline to 6 months
  change in LDL
Triglycerides | baseline to 6 months
  change in triglycerides
Glucose | baseline to 6 months
  change in glucose
Interleukin 6 (IL-6) | baseline to 6 months
  Change in IL-6
Interleukin 10 (IL-10) | baseline to 6 months
  change of IL-10 change in IL-10
C reactive protein (CRP) | baseline to 6 months
  change of CRP
Bone mineral density (BMD) | baseline to 6 months
  change in BMD
Body mass index (BMI) | Baseline to 6 months
  Change in BMI
Zinc levels | baseline to 6 months
  Change in zinc levels
Iron levels | baseline to 6 months
  Change in iron levels
A vitamin levels | baseline to 6 months
  change in A vitamin levels
C vitamin levels | baseline to 6 months
  change of C vitamin levels
D vitamin levels | baseline to 6 months
  change in D vitamin levels
E vitamin levels | baseline to 6 months
  change of E vitamin levels
Systolic blood pressure (SBP) | baseline to 6 months
  change in SBP
Diastolic blood pressure (DBP) | baseline to 6 months
  change in (DBP)